CLINICAL TRIAL: NCT00337948
Title: An Open-Labeled Pilot Study to Evaluate the Effects of High Dose PROCRIT (Epoetin Alfa) in Maintaining Hemoglobin Levels in Anemic Cancer Patients Receiving Chemotherapy on a Weekly or Every Four Week Regimen
Brief Title: An Efficacy and Safety Study of PROCRIT (Epoetin Alfa) in Cancer Patients Receiving Chemotherapy Every Week or Every Four Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004615
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-01

CONDITIONS: Chemotherapy; Anemia; Cancer
Keywords: Anemia; Epoetin Alfa; Chemotherapy; Anemia due to Cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of epoetin alfa at a starting dose of 60,000 Units (U) once every week (QW) to a target hemoglobin (Hb) of 12 g/dL (Initiation Phase), followed by a dose of 60,000 U once every other week (Q2W) to maintain a Hb range of 11.5 to 12.5 g/dL (Maintenance Phase) in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
Epoetin alfa administered three times weekly (150 U/kg) or once weekly (40,000 U) results in a response rate (defined as >= 2 g/dL hemoglobin (Hb) increase or Hb >= 12 g/dL) of approximately 65% of anemic chemotherapy patients and produces a mean hemoglobin rise of 1.8 g/dL. Higher weekly dosing may result in a higher response rate and a more timely mean hemoglobin rise while remaining safe. Additionally, limited data are available to show whether epoetin alfa maintenance therapy can be administered less frequently than weekly and still maintain hemoglobin levels. This is an open label, multicenter, non-randomized study to determine the safety and effectiveness of epoetin alfa given to cancer patients receiving chemotherapy every week or every four weeks.

Patients will receive up to 12 injections of epoetin alfa 60,000 U once every week (QW) subcutaneously (under the skin) for up to 12 weeks. Once a patient's hemoglobin level (Hg) has reached a target level of 12 g/dL, they will begin the Maintenance Phase. Patients who qualify for Maintenance Phase will receive up to 6 injections of 60,000 U every other week (Q2W) epoetin alfa under the skin for up to an additional 12 weeks to maintain hemoglobin 11.5 g/dL during chemotherapy administration. Doses will be held and adjusted downward if hemoglobin level rises to >13 g/dL or if a very rapid hemoglobin response occurs (e.g., an increase of more than 1.3 g/dL in a 2-week period).

Safety evaluations include clinical laboratory tests (hemoglobin and hematocrit), vital sign measurements (blood pressure), and incidence and severity of adverse events. In addition, the incidence of anti-erythropoietin antibodies at baseline and study completion/early withdrawal will be evaluated in patients who receive multiple doses of PROCRIT (Epoetin alfa). Patients will receive up to 12 injections of 60,000 U once every week (QW) epoetin alfa subcutaneously (under the skin) for up to 12 weeks. Once a patient's hemoglobin level (Hg) has reached a target level of 12 g/dL, they will begin the Maintenance Phase. Patients who qualify for Maintenance Phase will receive up to 6 injections of 60,000 U every other week (Q2W) epoetin alfa under the skin for up to an additional 12 weeks to maintain hemoglobin 11.5 g/dL during chemotherapy administration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy and receiving chemotherapy
* Baseline Hb of <= 11 g/dL
* Planned chemotherapy for a minimum of 16 weeks to be administered weekly or every 4 weeks
* Female patients with reproductive potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* No uncontrolled hypertension or recent history (within 6 months) of uncontrolled cardiac arrhythmias, pulmonary embolism, or thrombosis
* No transfusion of white blood cells or packed red blood cells within 28 days of Epoetin alfa treatment
* No prior treatment with Epoetin alfa or any other erythropoetic agent within the previous three months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-02; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving >= 2 g/dL Hb increase from baseline or Hb >= 12 g/dL in the Initiation Phase (up to 12 weeks).

SECONDARY OUTCOMES:
Proportion of patients with: >=1 g/dL Hb increase from baseline (up to 1.9 g/dL) in the Initiation Phase; those maintaining Hb level >11 g/dL (up to 11.4 g/dL); and those maintaining Hb level 11.5 to 12.5 g/dL in the Maintenance Phase (up to 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label Pilot Study to Evaluate the Effects of High Dose PROCRIT (Epoetin alfa) in Maintaining Hemoglobin Levels in Anemic Cancer Patients Receiving Chemotherapy on a Weekly or Every 4 Week Regimen. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=607&filename=CR004615_CSR.pdf